CLINICAL TRIAL: NCT02559648
Title: Evaluation of Efficacy of Denosumab in Patients With Thalassemia Major and Osteoporosis: A Randomized, Placebo-controlled, Single-site, Double Blind Phase 2b Clinical Trial
Brief Title: Denosumab vs Placebo in Patients With Thalassemia Major and Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ersi Voskaridou (Other)
Responsible Party: Sponsor-Investigator, Ersi Voskaridou, Director of National center of Thalassaemia and Haemoglobinopathies of Laikon General Hospital of Athens, Laikο General Hospital, Athens
Organization: Laikο General Hospital, Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EL-THOS-001; 2014-000931-18 (EudraCT Number)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Thalassemia Major; Osteoporosis
MeSH Terms: conditions — beta-Thalassemia; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Active Comparator): In Group A, 60 mg Denosumab will be administered sc, every 6 months for 12 months for a total of 2 doses (day 0 and day 180)
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): In Group B placebo will be administered sc, every 6 months for 12 months for a total of 2 doses (day 0 and day 180)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — Patients will be randomly assigned, in a 1:1 fashion, to the two therapeutic arms (Group A, Group B, respectively), upon enrollment in the study.
  The effect of denosumab on lumbar spine BMD (bone mineral density) in patients with Thalassemia Major and Osteoporosis as compared with control at 12 months will be evaluated.
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo — Patients will be randomly assigned, in a 1:1 fashion, to the two therapeutic arms (Group A, Group B, respectively), upon enrollment in the study.
  The effect of denosumab on lumbar spine BMD (bone mineral density) in patients with Thalassemia Major and Osteoporosis as compared with control at 12 months will be evaluated.
  Arms: Placebo

SUMMARY:
This is a single-site, randomized, placebo-controlled, double blind phase 2b clinical trial. Patients with Thalassemia will participate in this study and will be treated with Denosumab or placebo. The effect of Denosumab on lumbar spine BMD in patients with Thalassemia Major and Osteoporosis will be evaluated as compared with control (placebo) at 12 months.

DETAILED DESCRIPTION:
This is a single-site, randomized, placebo-controlled, double blind phase 2b clinical trial. Patients with Thalassemia and Bone Mass Density (BMD) T-score between -2.5 and - 4.0 in at least one of the examined sites will participate in this study and will be treated with Denosumab or placebo.

Patients will be assigned into two (2) treatment groups:

* In Group A, 60 mg Denosumab will be administered sc, every 6 months for 12 months for a total of 2 doses (day 0 and day 180).
* In Group B placebo will be administered sc, every 6 months for 12 months for a total of 2 doses (day 0 and day 180) (Appendix I and Appendix II).

Patients will be randomly assigned, in a 1:1 fashion, to the two therapeutic arms (Group A, Group B, respectively), upon enrollment in the study.

The effect of Denosumab on lumbar spine BMD (bone mineral density) in patients with Thalassemia Major and Osteoporosis as compared with control at 12 months will be evaluated. Also the effect on femoral neck and wrist bone BMD, on markers of bone remodeling and the safety profile will be evaluated as well. All subjects will receive a subcutaneous injection of Denosumab or placebo administered by a health care professional on days 0 and 180 (±3).

ELIGIBILITY:
Inclusion Criteria:

* Adults (>30 years of age) described as skeletally mature subjects
* Thalassemia Major
* Low BMD (T-score <-2.5) in one of the 3 studied sites (lumbar spine, femoral neck, wrist).
* Have signed the informed consent form (consent should be taken before any study-specific procedure is performed).

Exclusion Criteria:

* BMD T-score < -4.0 in one of the 2 studied sites (lumbar spine, femoral neck).
* Previous administration of denosumab from clinical trials or others (e.g. commercial use).
* Current participation in another clinical trial or having received any investigational product within the last 3 months.
* Impaired renal function as determined by an estimated glomerular filtration rate (eGFR) of ≤ 30 mL/min (using the Chronic Kidney Disease-Epidemiology, ((CKD-EPI) formula).
* Patients with sickle cell disease.
* Known to have a liver failure or chronic hepatic disease e.g. cirrhosis, chronic hepatitis; or elevated transaminases defined as Alanine Transaminase (ALT) and/or Aspartate Transaminase (AST) > 2 fold the upper limit of normal laboratory range.
* Heart failure (NYHA above 2).
* Patients with life expectancy of less than one year.
* Subject refuses to use a reliable contraceptive method (oral contraceptives, progesterone implants, intrauterine device, condoms) throughout the study by women of childbearing potential. Women of childbearing potential agree to use 2 highly effective forms of contraception and to continue this practice for 7 months after last injection of study medication.
* Pregnancy, planning a pregnancy or currently lactating
* Severe concurrent illness which in the investigator's opinion may confound patient evaluation, e.g. malignancy (except basal cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years.
* Known alcohol or drug abuse or any other condition associated with poor compliance
* Patients that have received oral bisphosphonates within 6 months of study enrollment or intravenous bisphosphonates, fluoride and strontium ranelate within 1 year of study enrollment.
* Parathormone (PTH), PTH derivatives, teriparatide, odanacatib, anabolic steroids, testosterone, glucocorticosteroids (> 5 mg/day of prednisone equivalent for > 10 days), systemic hormone-replacement therapy, selective estrogen receptor modulators (SERMs), raloxifene, tibolone, calcitonin or calcitriol use within the last 6 weeks.
* Evidence of hyper- or hypothyroidism; patients with an abnormal Thyroid stimulating hormone (TSH) level on thyroid treatment (patients on stable thyroid treatment with a normal TSH allowed); current hyper- or hypoparathyroidism; current hyper or hypocalcemia (hypocalcemia based on albumin adjusted serum calcium < 8.5 mg/dL); vitamin D deficiency (25-hydroxy Vitamin D level < 12 ng/mL; if repeat 12-20 ng/mL after repletion, subject will be allowed); rheumatoid arthritis; Paget's disease; bone disease that would interfere with interpretation of findings.
* Known sensitivity to mammalian cell-derived drug products.
* History of any Solid Organ or Bone Marrow Transplant
* History of osteonecrosis of the jaw, and/or recent tooth extraction or other dental surgery; or planned invasive dental work during the study.
* Intolerance to calcium supplements.
* Malabsorption syndrome; severe malabsorption including Celiac disease, Short Bowel Syndrome, Crohn's disease, Previous Gastric Bypass.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The percent change in the lumbar spine BMD | 12 months
  The primary objective is to evaluate the effect of Denosumab (plus vitamin D & calcium) on lumbar spine BMD in patients with Thalassemia Major and Osteoporosis as compared with control (placebo plus vitamin D & calcium) at 12 months

SECONDARY OUTCOMES:
The percent change in BMD of the total hip and femoral neck | 12 months
  To evaluate the effect of Denosumab (plus vitamin D & calcium) on femoral neck and wrist bone BMD in patients with Thalassemia Major and Osteoporosis as compared with control (placebo plus vitamin D & calcium) at 12 months
The percent change in BMD at the distal third radius | 12 months
  To evaluate the effect of Denosumab (plus vitamin D & calcium) on femoral neck and wrist bone BMD in patients with Thalassemia Major and Osteoporosis as compared with control (placebo plus vitamin D & calcium) at 12 months
The percent change in serum C-Termina Telopeptide (sCTX) at Month 3 post injection | 3 months
  To evaluate the effect of Denosumab on markers of bone remodeling of patients with Thalassemia Major and Osteoporosis.

OTHER OUTCOMES:
Adverse event incidence by system organ class and preferred term | 12 months
  Seventeen cases of adverse events were reported. 14/17 were classified as mild(grade 1). 3/14 mild adverse eents concerned the placebo group. 11/14 of the mild adverse events concerned abnormalities of blood or biochemical testing. Only 3 of them had headache, diarrhea and fever. Three serious adverse events in denosumab group were pleural effusion(grade 3), supraventricular tachycardia(grade 4) and atrial fibrillation (grade3). These all three events were defined as unrelated to study drug.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  To evaluate the safety profile of Denosumab in patients with Thalassemia Major and Osteoporosis.
  Hematological parameters: Hemoglobin (Hb), White blood cell number (WBC) and platelets number
  Biochemical parameters: ALT U/L, AST U/L, Alkaline phosphatase IU/L, CPK IU/L, Calcium mg/dL, Creatinine mg/dL, Direct bilirubin mg/dL, LDH U/L, Phosphate mg/dL, Total bilirubin mg/dL, Total protein g/dL, Urea mg/dL, Uric acid mg/dL, albumin g/dL, ferritin ng/mL, glucose mg/dL, iron μg/dL, magnesium mg/dL, potassium mEq/L, sodium mEq/L, γGT IU/L.
Changes in general appearance at each visit | 12 months
  General appearance of the patients will be assessed at each visit as "normal" of "affected".
Changes in skin contour at each visit | 12 months
  At each visit all patients will be evaluated for potential changes in skin contour and will be classified as i) normal or pale and ii) icteric or non-icteric
Changes in cardiology clinical examination at each visit | 12 months
  At each visit all patients will be evaluated for potential changes in heart clinical examination assessed by auscultation that will be classified as normal or abnormal
Changes in ECG at each visit | 12 months
  At each visit all patients will be evaluated for ECG changes regarding the cardiac rhythm, the cardiac rate, the P Wave, the PR Interval, the QRS Complex, the QT Interval, and will be classified as normal or abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Ersi Voskaridou, Doctor, Principal Investigator — General Hospital of Athens "Laikon"
Locations (1):
- General Hospital of Athens "Laikon", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voskaridou E, Ntanasis-Stathopoulos I, Papaefstathiou A, Christoulas D, Dimopoulou M, Repa K, Papatheodorou A, Peppa M, Terpos E. Denosumab in transfusion-dependent thalassemia osteoporosis: a randomized, placebo-controlled, double-blind phase 2b clinical trial. Blood Adv. 2018 Nov 13;2(21):2837-2847. doi: 10.1182/bloodadvances.2018023085. PMID 30381400